CLINICAL TRIAL: NCT00892255
Title: Microwave Ablation of Resectable Liver Tumors
Status: Withdrawn | Type: Observational
Sponsor: St. Joseph Hospital of Orange (Other)
Responsible Party: Sponsor
Other Study IDs: 09-008 Microwave Ablation
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: Liver cancer; Tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Microwave Ablation — Tumor tissue from the liver is inter-operatively treated with the microwave ablation device to measure the destruction of tissue.

SUMMARY:
The purpose of this protocol is to pathologically evaluate the destruction by microwave ablation of primary and metastatic liver tumors. The primary aim is to measure tissue destruction with the MedWaves Microwave Ablation/ Coagulation Ablation System.

DETAILED DESCRIPTION:
Minimally invasive surgical alternatives are becoming more attractive for the treatment of malignancy.The goal is to reduce morbidity and mortality and increase the ability to treat patients in the outpatient setting. Image-guided ablation is becoming an attractive alternative because of its relative low cost, its ability to provide large regions of coagulative necrosis in a controlled fashion, and its relatively low toxicity. Although image-guided ablative techniques have been extensively investigated for the treatment of liver tumors, there has been limited experience with microwave ablation (MWA) in the liver. This study will evaluate the treatment effect of MWA in liver tumors. Patients undergoing planned surgical removal of liver tumors will have the tumors intra-operatively treated with MWA. The histological changes will be evaluated upon removal of the specimen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary or metastatic liver cancer for which surgery is planned
* All participants need to be fully able to give informed consent

Exclusion Criteria:

* Mental or legal incompetence
* Impaired decision-making capacity
* Pregnant women may not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for liver resection, either for primary or metastatic disease
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Measure of the tissue destruction with the MedWaves Microwave Ablation/ Coagulation Ablation System | 30 Days
  Measure of the tissue destruction with the MedWaves Microwave Ablation/ Coagulation

CONTACTS AND LOCATIONS:
Overall Officials: Hisham El-Bayar, MD, Principal Investigator — St. Joseph Hospital of Orange
Locations (1):
- The Center for Cancer Prevention & Treatment at St. Joseph Hospital, Orange, California, United States